CLINICAL TRIAL: NCT07321938
Title: Accuracy Evaluation of the Owlet OSS 3.0-M1 Sensor in Toddlers and Preschoolers
Acronym: TOPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Owlet Baby Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OWL-TOP-2501
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: pulse oximetry; pediatrics; Owlet

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Owlet OSS 3.0-M1 Sensor (Experimental): Owlet OSS 3.0-M1 Sensor accuracy evaluation compared to a reference pulse oximeter.
  Interventions: Device: Application and monitoring with an Owlet OSS 3.0-M1 Sensor; Device: Reference Pulse Oximeter

INTERVENTIONS:
Device: Application and monitoring with an Owlet OSS 3.0-M1 Sensor — Owlet OSS 3.0-M1 Sensor
Device: Reference Pulse Oximeter — Application and monitoring with an FDA cleared reference pulse oximeter

SUMMARY:
The purpose of the study is to collect information from the Owlet OSS 3.0-M1 Sensor in toddlers and preschoolers to evaluate accuracy.

DETAILED DESCRIPTION:
The objective of this study is to collect evidence to verify the accuracy of the Owlet OSS 3.0-M1 Sensor to measure SpO2 and pulse rate in children 19-60 months in a simulated use environment as compared to an FDA cleared reference pulse oximeter.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 19 months and ≤ 60 months of age.
2. Subject's current body weight is ≥ 6 lbs.
3. Subject/legal guardian is fluent in both written and spoken English.
4. Subject is willing and able to follow study requirements
5. Legal guardian has provided consent.

Exclusion Criteria:

1. Subject has preexisting cardiovascular or respiratory disease or conditions.
2. Subjects with abnormalities (e.g., limb deformities, open wounds, severe edema) at the planned application sites that would interfere with system measurements.
3. The device(s) are unable to fit properly without risk of injury (e.g., hook of VELCRO is against the skin, wrap is too tight and constricting).
4. Subject has skin irritation at the location of device placement.
5. Subject has known allergies to adhesive.

Ages: 19 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Pulse rate accuracy | 2 hours
  Average root mean square (ARMS) error between the pulse rate measured by the Owlet OSS 3.0-M1 vs. a reference pulse oximeter
SpO2 Accuracy | 2 hours
  The average root mean square difference between the Owlet OSS 3.0-M1 Sensor vs. readints from an FDA cleared reference pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Stratmann, MD, PhD, Principal Investigator — Vital Signs Research Group, LLC
Locations (1):
- Vital Signs Research Group, LLC, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data collected during the course of this study are specifically intended for a regulatory submission and may or may not be shared publicly.